CLINICAL TRIAL: NCT01693302
Title: Timing of Meal Insulin Boluses to Achieve Optimal Postprandial Glycemic Control in Patients With Type 1 Diabetes
Brief Title: Timing of Meal Insulin Boluses for Optimal Postprandial Glycemic Control in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 06-0994
Record Dates: First submitted 2009-09-09; First posted 2012-09-26 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Type 1 Diabetes
Keywords: Blood Glucose; Meal insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- -20 minute insulin (Experimental): Insulin for the meal is given 20 minutes prior to starting the meal.
  Interventions: Other: Insulin
- 0 minute insulin (Experimental): Insulin for the meal is given immediately before starting to eat.
  Interventions: Other: Insulin
- +20 minute insulin (Experimental): Insulin is given 20 minutes after the start of the meal.
  Interventions: Other: Insulin

INTERVENTIONS:
Other: Insulin — The timing of insulin delivery varies with each study visit. The dose is given based on carbohydrate content and blood glucose level. The insulin is given either 20 minutes before the meal, immediately before the meal, or 20 minutes after the meal.
  Other Names: Insulin time

SUMMARY:
Blood glucose levels in patients with type 1 diabetes tend to peak after eating a meal due to the delayed action of insulin when compared to carbohydrate absorption from food. It is the hypothesis of the investigator that administering the insulin for a meal 20 minutes before the meal will result in lower blood glucose peaks compared to administration of insulin immediately before or 20 minutes after starting to eat.

All subjects will eat the same meal on three different occasions. Insulin will be administered at one of the three times at each visit.

DETAILED DESCRIPTION:
Subjects enrolled in this study will be between the ages of 12 and 30 years inclusive. All subjects will be on an insulin pump and use carbohydrate counting as their method for insulin dosing at a meal.

Subjects in this study will complete three study visits lasting from approximately 8:30am until 1:30pm. At each visit, the subject will eat the same frozen breakfast meal. Subjects will be supplied with the same insulin to maintain consistency between visits and between subjects.

Insulin will be administered at different times, depending upon the randomization group assigned to the participant. The three different times the insulin will be given is either 20 minutes before the meal, immediately before the meal and 20 minutes after the meal. All subjects will complete all three insulin bolus times. Blood glucose will be measured by fingerstick every 30 minutes until the completion of the visit.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 30 years of age, inclusive
* Clinical diagnosis of T1D and using daily insulin therapy for at least 1 year
* Using carbohydrate counting to dose meal time insulin
* HbA1c value upon enrollment greater than 6.0% and less than 12.0%
* Using CSII therapy for diabetes management for at least three months
* Able and willing to give informed consent/assent to participate
* No expectation that the subject will be moving out of the area of the clinical center during the study
* Willing to consume the same standard frozen meal on all three visits

Exclusion Criteria:

* The presence of a significant medical disorder that in the judgment of the investigator will affect the wearing of the CGMS sensors or the completion of any aspect of the protocol
* Being unable or unwilling to give informed consent
* Having documented hypoglycemia unawareness
* An episode of severe hypoglycemia (seizure or loss of consciousness) or of ketoacidosis in the past six months

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2007-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Blood glucose area under the curve | 9:00am until 1:30pm

SECONDARY OUTCOMES:
Glucose values one hour after the meal | 10:30am
Glucose values two hours after the beginning of the meal | 11:30am

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chase, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Barbara Davis Center, Aurora, Colorado, United States